CLINICAL TRIAL: NCT05827367
Title: High-power Pain Thershold Ultrasound Versus Myofascial Release in Patients With Chronic Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Menna Ali mohammed tolba, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPPTUS versus MFR IN PF
Record Dates: First submitted 2023-02-27; First posted 2023-04-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Plantar Fascitis
Keywords: high power pain thershold ultrasound; Planter fasciitis; Myofascial release
MeSH Terms: interventions — Ultrasonography; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high power pain thershold ultrasound (Experimental): Patients will reseiv high power pain ultrasound
  ,intrinsic muscle strength and plantar fascia streatching
  Interventions: Device: Ultrasound; Other: Strength and stretching
- myofascial release (Experimental): Plantar fascia myofascial release,gastrocnmias Myofascial release ,soluse myofascial release,foot interstice muscle strength and plantar fascia streatching
  Interventions: Other: Myofascial release technique; Other: Strength and stretching
- control arm (Placebo Comparator): Plantar fascia stretching and foot interstice muscle strength
  Interventions: Other: Strength and stretching

INTERVENTIONS:
Device: Ultrasound — The high-power pain threshold ultrasound (HPPTUS) In this technique, "which be applied in continuous mode with intensity from t0.5 to 2 watt/cm to elicit pain threshold the US probe was kept motionless, and the intensity progressively increased until the maximum level of pain patient can endure was selected, it was maintained on this level for 3 to 4 seconds and then decreased to half intensity for 15 seconds the treatment process was repeated three times.
  Arms: high power pain thershold ultrasound
Other: Myofascial release technique — Plantar fascia myofascial release Soluse muscle myofascial release Gastrocnmias muscle myofascial release
  Arms: myofascial release
Other: Strength and stretching — Plantar fascia stretching Interstice foot muscles strengthing

SUMMARY:
1. To compare effect of high power pain threshold ultrasound versus myofascial release technique on pain pressure threshold over the medial calcaneal tuberosity of the involved heel in treating of chronic planter fasciitis patients
2. To compare effect of high power pain threshold ultrasound versus myofascial release technique on pain intensity in treating of chronic planter fasciitis patients.
3. To compare effect of high power pain threshold ultrasound versus myofascial release technique on ankle disability function in treating of chronic planter fasciitis patients.
4. To compare effect of high power pain threshold ultrasound versus myofascial release technique on ankle active dorsiflexion range of motionin treating of chronic planter fasciitis patients.
5. To compare effect of high power pain threshold ultrasound versus myofascial release technique on walk endurance. In treating of chronic planter fasciitis patients.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is The most common cause of plantar heel pain(PHP) is a degeneration of the plantar fascia as a result of repetitive micro tears of the fascia that lead to an inflammatory reaction, and is not a primary inflammatory process that most believe it to be the cause of plantar fasciitis is unknown but is believed to be multifactorial, with abnormal biomechanics. It is the most common cause of heel pain about 4% to 7% of the population suffer from it. There are many risk factors for plantar fasciitis include excessive foot pronation or flat feet (pesplanus), high arches (pescavus), tight Achilles tendon or gastrocnemius muscle (equinus), tight intrinsic foot muscles, limb length discrepancy, obesity, running, prolonged standing or walking, poor-fitting shoes, and improper gait. Many patients complain of heel pain in the morning or after rising from prolonged sitting, with relief upon initiation of movement. Physical examination will reveal pain to palpation of the medial plantar calcaneal region, pain with dorsiflexion, and tightness of the Achilles tendon or the gastrocnemius muscle ,.

Plantar heel pain is associated with impaired health-related quality of life including social isolation, a poor perception of health status and reduced functional capabilities.

The high-power pain threshold ultrasound (HPPTUS) technique is one of the therapeutic ultrasound modifications used to treat myofascial pain syndrome.

HPPTUS is considered as an effective treatment for Myofascial pain syndrome which be applied in continuous mode with intensity from 0.5 to 2 watt/cm to elicit pain threshold the US probe was kept motionless, and the intensity progressively increased until the maximum level of pain patient can endure was selected, it was maintained on this level for 3 to 4 seconds and then decreased to half intensity for 15 seconds the treatment process was repeated three times.

performed clinical study to compare (HPPTUS) technique with the traditional ultrasound technique in patients with myofascial pain syndrome. The results showed that HPPTUS was much more effective than the traditional technique, pain reduction and improvement of range of motion (ROM) were significant in a smaller number of sessions.

Myofascial release (MFR) is the application of a low load, long duration stretch to the myofascial complex, intended to restore optimal length, decrease pain, and improve function .MFR effect on (PF) by decreasing in tension over the plantar fascia and decrease of risk factors, such as tightness of the gastrocnemii and soleus muscles and restricted ankle dorsiflexion Several treatment methods are available to relieve symptoms associated with plantar fasciitis. These include stretching, manual therapy, dry needling, shockwave therapy, physical agents (electrotherapy, low-level laser therapy, phonophoresis, and ultrasound), lifestyle counseling, anti-inflammatory injections, and mechanical treatments such as taping, rocker shoes, and ankle-foot orthoses including night splints. Mechanical treatments are promising due to the low risk of complications, good accessibility, and high capacity to relieve the mechanical load on the plantar fascia during functional tasks of daily life. The effectiveness of mechanical treatment on plantar fasciitis has previously been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of plantar fasciitis more than three months ago
* Patient's age ranged between 40-60 years old
* Patients with body mass index (MBI)<30kg/m2

Exclusion Criteria:

* Patients with any prior surgery to distal tibia, fibula, ankle joint or rear foot region.
* presence of any red flags i.e., tumor, fracture, and heterotrophic ossification and had acute inflammatory condition at ankle-foot region were excluded from the study.
* Deformity of foot and ankle complex and subjects with referred pain due to sciatica and other neurological disorders

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
pain pressure threshold | Change at pain pressure thershold through 4 weeks
  pain pressure threshold over the medial calcaneal tuberosity of the involved heel will be measured by pressure algometer.

SECONDARY OUTCOMES:
Pain intensity at first step after prolonged setting | Change at pain intensity through 4 weeks
  Pain intensity at first step after prolonged setting will be measured by numerical pain rating scale it rang from 0 that means no pain and 10 that means the worst pain ever

OTHER OUTCOMES:
Disability function of ankle joint | Change at disability function of ankle through 4 weeks
  Disability function of ankle joint will be measured by Arabic version of foot function index scale.that consist of 23 question each one score range from 0 it mean no pain to 10 that means worst pain
Ankle joint dorsi flexion | Change at ankle dorsi flexion through 4 weeks
  Ankle joint dorsi flexion will be measured by manual goniometer
Walk endurance | Change at walk endurance through 4 weeks
  Walk endurance will be measured by 6-min walk test

CONTACTS AND LOCATIONS:
Overall Officials: doaa rafat, Lecturer, Study Director — Cairo University; amaal hassan, Professor, Study Director — Cairo University; mohammed kaddah, Professor, Study Director — Cairo University